CLINICAL TRIAL: NCT01689870
Title: Phase 1/2 Study of the Combination of a Mouse Monoclonal Antibody to OX40 and Ipilimumab in Patients With Metastatic Melanoma
Brief Title: Study of the Combination of Anti-OX40 and Ipilimumab in Patients With Metastatic Melanoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: AgonOx (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUD2012-005
Record Dates: First submitted 2012-09-18; First posted 2012-09-21 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Metastatic Melanoma
Keywords: OX40; Anti-OX40; Ipilimumab; Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phase 1 Cohort 1 (Experimental): Ipilimumab will be administered at 3 mg/kg i.v. over 90 minutes every 3 weeks for a total of 4 doses, starting on Day 1. Anti-OX40 will be administered at 0.1 mg/kg over 60 minutes only in the first week on Days 1, 3 and 5.
  Interventions: Drug: Anti-OX40; Drug: Ipilimumab
- Phase 1 Cohort 2 (Experimental): Ipilimumab will be administered at 3 mg/kg i.v. over 90 minutes every 3 weeks for a total of 4 doses, starting on Day 1. Anti-OX40 will be administered at 0.2 mg/kg over 60 minutes only in the first week on Days 1, 3 and 5.
  Interventions: Drug: Anti-OX40; Drug: Ipilimumab
- Phase 1 Cohort 3 (Experimental): Ipilimumab will be administered at 3 mg/kg i.v. over 90 minutes every 3 weeks for a total of 4 doses, starting on Day 1. Anti-OX40 will be administered at 0.4 mg/kg over 60 minutes only in the first week on Days 1, 3 and 5.
  Interventions: Drug: Anti-OX40; Drug: Ipilimumab
- Phase 2 Cohort 4 (Experimental): Ipilimumab will be administered at 3 mg/kg i.v. over 90 minutes every 3 weeks for a total of 4 doses, starting on Day 1. Anti-OX40 will be administered i.v. at the Phase 1 Maximum Tolerated Dose over 60 minutes only in the first week on Days 1, 3 and 5.
  Interventions: Drug: Anti-OX40; Drug: Ipilimumab

INTERVENTIONS:
Drug: Anti-OX40 — Anti-OX40 will be administered i.v. over 60 minutes only in the first week on Days 1, 3 and 5
  Other Names: CD134 mab
Drug: Ipilimumab — Ipilimumab will be administered at 3 mg/kg i.v. over 90 minutes every 3 weeks for a total of 4 doses, starting on Day 1
  Other Names: YERVOY

SUMMARY:
This is an open label, two-phase study combining a dose escalation Phase 1 with a proof-of-concept Phase 2 in patients with unresectable or metastatic melanoma, for whom treatment with ipilimumab is indicated.

The purpose of the Phase 1 is to determine the Anti-OX40 Maximum Tolerated Dose (MTD) and the secondary objectives are anti-OX40 pharmacokinetics, biological activity and the tumor response assessed by the Immune-related Response Criteria.

The purpose of Phase 2 is to determine tumor response (by irRC) and the secondary objectives are anti-OX40 pharmacokinetics, biological activity and Safety/Tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable or metastatic melanoma, for whom treatment with Ipilimumab is indicated
* Radiologically measurable disease by immune-related Response Criteria
* ECOG performance status of 0-1.
* Anticipated lifespan greater than 12 weeks.
* At the time of day 1 of the study, patients must be at least 3 weeks since surgery
* At the time of day 1 of the study, patients with brain metastases must be asymptomatic and, at least 8 weeks without tumor progression after any whole brain radiotherapy, at least 4 weeks since craniotomy and resection or stereotactic radiosurgery, at least 3 weeks without new brain metastases as evidenced by MRI/CT
* The following laboratory parameters must be within the ranges specified: Hemoglobin-≥ 9 g/dL, WBC-≥ 3.0 x 109/L, INR-≤ 1.5, Total Bilirubin-≤ 1.9 g/dL & AST/ALT-≤ 3 x ULN
* Have been informed of other treatment options.
* At least 18 years. Able and willing to give valid written informed consent.

Exclusion Criteria:

* Any contraindications for ipilimumab/Yervoy®.
* Prior exposure to ipilimumab/Yervoy®
* Prior exposure to Anti-OX40 or a mouse monoclonal antibody.
* History of severe allergic reactions to any unknown allergens or anti-OX40 Autoimmune disease except for autoimmune thyroiditis or vitiligo.
* Unresolved immune related adverse events following prior biological therapy.
* Metastatic disease to the central nervous system for which other therapeutic options, including radiotherapy, may be available.
* Known immunodeficiency or HIV, Hepatitis B or Hepatitis C positivity.
* Other serious illnesses (e.g., serious infections requiring antibiotics).
* Participation in any other clinical trial involving another investigational agent within 4 weeks prior to day 1 of the study.
* Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study.
* Lack of availability for immunological and clinical follow-up assessments.
* Women who are breast feeding or pregnant as evidenced by positive serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) done within 72 hours of first dosing.
* Women of childbearing potential not using a medically acceptable means of contraception for the duration of the study.
* Any condition that, in the clinical judgment of the treating physician, is likely to prevent the patient from complying with any aspect of the protocol or that may put the patient at unacceptable risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Assess safety and tolerability according to the National Cancer Institute CTCAE v4.0 (Phase 1 and 2) | Up to 16 weeks
  Laboratory tests, vital sign measurements, physical exams and patient interviews will be performed to detect new abnormalities and deteriorations of any pre-existing conditions
Assess Tumor Response by the Immune-related Response Criteria (Phase 2) | Baseline, Week 12 & week 16
  Tumor Response by irRC is defined as irPR or irCR over a period of at least 4 weeks

SECONDARY OUTCOMES:
Determine Anti-OX40 serum concentrations | Baseline, on days 1, 3 & 5 30 minutes after Anti-OX40 end of infusion, and on days 8 and 15
  The serum concentration of Anti-OX40 (CD134) will be determined from its binding to OX40 as measured by ELISA
Assess the biological activity of anti-OX40 in combination with ipilimumab | Baseline, Day1, day 3, day 5 day8, day 15, day 22 day 43, day 64, day 85 & 113
  The biological activity of anti-OX40 in combination with ipilimumab will be assessed by:
  * Determining immunologic changes in the tumor microenvironment by characterization of tumor-infiltrating lymphocytes (TILs), assessment of antigen-specific T cell responses and immunohistochemical (IHC) characterization of tumor and peri-tumoral tissue
  * Characterizing circulating T-cell subsets by flow cytometry
  * Assessing antigen specific immune responses by ELISA
  * Characterizing surface markers on lymphocytes and peripheral blood cells by flow cytometry
  * Measuring serum level of soluble factors (cytokine profiling)
  * mRNA/miRNA profiling to analyse gene transcription and/or miRNA expression

CONTACTS AND LOCATIONS:
Overall Officials: Jedd Wolchok, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Brendan D Curti, MD, Principal Investigator — Providence Health & Services